CLINICAL TRIAL: NCT00799279
Title: Comparative Evaluation of the Efficacy and Cost-effectiveness of Two Interventions for Integrating Smoking Cessation Into Routine Primary Care Practice: A Cluster-randomized Trial
Brief Title: Integrating Smoking Cessation Into Routine Primary Care Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other); Canadian Tobacco Control Research Initiative (Other)
Responsible Party: Paul McDonald, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15053; CTCRI 019826 (Other Grant/Funding Number: Canadian Tobacco Control Research Initiative); CTCRI 19813 (Other Grant/Funding Number: Canadian Tobacco Control Research Initiative)
Record Dates: First submitted 2008-11-17; First posted 2008-11-27 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Smoking Cessation
Keywords: smoking; cessation; family medicine; evidence-based; knowledge translation; smoking cessation, primary care
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up Counseling Arm (Experimental): smoking cessation training for providers,practice tools for providers, patient quit plan, and follow-up telephone counselling for smokers
  Interventions: Behavioral: Smoking cessation training, support, and telephone follow-up
- Practice Support Arm (Active Comparator): smoking cessation training for providers,practice tools for providers, patient quit plan for smokers.
  Interventions: Behavioral: smoking cessation intervention

INTERVENTIONS:
Behavioral: Smoking cessation training, support, and telephone follow-up — The CF group will receive the same smoking cessation training and practice support tools delivered to the PS group. In addition, patients in the FC group who are smokers and are willing to set a quit date within the next 30 days and who have set a quit date will be enrolled in an interactive voice response (IVR)-mediated telephone follow-up and counselling system. The IVR system will automatically contact patients via telephone 7 days before their TQD, and 5, 14, 30, and 60 days after their TQD to check the patients' smoking status, potential concerns, and their risk of relapse.
  Arms: Follow-up Counseling Arm
Behavioral: smoking cessation intervention — Intervention practices will be provided with training in smoking cessation, and will be supported with integrating a waiting room screener for smoking and smoking consult form and patient quit plan into their practice routines.
  Arms: Practice Support Arm

SUMMARY:
The aim of this study is to determine if providing smokers identified in family doctors offices with follow-up counselling enhances their success with quitting and the number of health professionals helping patients with quitting. Six to eight family medicine clinics will be involved in the study. We will compare the frequency of addressing smoking with patients and the proportion of smokers who are successful with quitting 16-weeks following the clinic appointment between practices. It is hypothesized that the addition of follow-up counseling to a multi-component smoking cessation intervention will improve smoking outcomes.

DETAILED DESCRIPTION:
A family doctor's advice to quit has been shown to increase a smoker's motivation to quit. Despite the evidence supporting the importance of smoking cessation, there is a well-documented practice gap in the rates at which smoking cessation is being addressed by practitioners. The primary objectives of this research study are to determine whether adjunct telephone-based smoking cessation follow-up counselling when delivered as part of a multi-component intervention:

1. Increases the rate at which evidence-based smoking cessation interventions are delivered to smokers identified in family doctors offices, compared to providing only practice supports.
2. Increases smoking abstinence as measured three months after the estimated target quit date (i.e.16 weeks) compared to providing only practice supports.
3. Is more cost-effective (cost/quit) than providing only practice supports to family doctors offices.

A two-arm before-after matched-pair cluster randomized trial, will test the effectiveness of two strategies for integrating smoking cessation treatments into primary care practice routines and enhancing cessation. Six to eight family doctors offices will be randomized to either a practice support (PS) group, or a follow-up counseling (FC) group. From each of the intervention practices a cross-sectional sample of 50 eligible smokers will be recruited pre- and post-intervention to assess 5A's delivery and smoking abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Practices will be eligible for participation in the present study if they meet the following criteria:

  1. Practice is a family health team (FHT), family health group (FHG); or family health network (FHN);
  2. All physicians within the practice are willing to participate in the study;
  3. Practice will see an average of 50 patients per day and 10% of patients are smokers;
  4. Practice is willing to provide consent to contact patients in waiting rooms and survey patients during office hours and by telephone.
* Patients will be eligible to participate in the study if they meet the following criteria:

  1. Patient is seen in clinic for annual exam or non-urgent visit;
  2. Patient is a current smoker (>1 cigarette per day on most days of the week);
  3. Patient is 18 years of age or older;
  4. Patient is able to read and understand English or French;
  5. Patient has a home or mobile telephone which can be used to receive follow-up telephone counselling calls

Exclusion Criteria:

* Patients who do not have the mental capacity to provide informed consent and complete study protocols will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
smoking abstinence | 16-weeks
  Self-report and biochemically validated point prevelence smoking abstinence

SECONDARY OUTCOMES:
cost-effectiveness | 16-weeks
Rate of provider delivery of evidence-based smoking treatments | exit survey on day of clinic visits
  Rates of providers, asking, advising, assessing, assisting, and arranging were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Paul McDonald, PhD, Principal Investigator — University of Waterloo